CLINICAL TRIAL: NCT00292006
Title: The Efficiency of Computerized Tomography to Aid in the Diagnosis of Pediatrics Scaphoid Fractures
Brief Title: Computerized Tomography to Help Diagnosis Pediatrics Scaphoid Fractures.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11955
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2006-02

CONDITIONS: Scaphoid Bone; Fracture
Keywords: clinical scaphoid fracture; pediatric
MeSH Terms: conditions — Fractures, Bone | interventions — Tomography, X-Ray Computed

INTERVENTIONS:
Device: Computerized tomography

SUMMARY:
The purpose of this study is to find out whether computerized tomography will be better than plain radiographs in determining pediatrics scaphoid fractures.

DETAILED DESCRIPTION:
Background: The use of plain radiograph in the detection of pediatrics scaphoid fractures has low specificity and sensitivity. Patients with documented anatomical snuffbox tenderness and negative plain radiographs are casted in thumb spica casts and seen by a pediatrics orthopedics surgeon. However few patients with clinical scaphoid fractures have documented scaphoid fractures, with the most common injury of soft tissue injury to the surrounding tissues. The use of CT scan to detect scaphoid fractures is not well documented and may be an appropriate substitute for plain radiographs.

Hypothesis: CT scan of the wrist will have higher sensitivity and specificity in detecting pediatrics scaphoid fracture than plain radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Pain in anatomical snuffbox, Negative radiographs, less than 18 years old, older than 6 years old, injury less than 1 week old and provision of informed consent

Exclusion Criteria:

* Previous injury to scaphoid bone, other injuries on the same extremity, vascular injury present at the injury site, fracture seen on initial radiographs, injury >1 week old, inability for patient to comply with rehabilitation or form completion, likely problems in maintaining patient follow-up

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2007-06

PRIMARY OUTCOMES:
Fracture diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Tim P Carey, MD, FRCSC, Study Chair — Western University, Canada
Locations (1):
- London Health Sciences Center Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Temple CL, Ross DC, Bennett JD, Garvin GJ, King GJ, Faber KJ. Comparison of sagittal computed tomography and plain film radiography in a scaphoid fracture model. J Hand Surg Am. 2005 May;30(3):534-42. doi: 10.1016/j.jhsa.2005.01.001. PMID 15925164
- [Background] Breederveld RS, Tuinebreijer WE. Investigation of computed tomographic scan concurrent criterion validity in doubtful scaphoid fracture of the wrist. J Trauma. 2004 Oct;57(4):851-4. doi: 10.1097/01.ta.0000124278.29127.42. PMID 15514541